CLINICAL TRIAL: NCT03512041
Title: Effect of Number of Remote Limb Ischemic Conditioning Cycles on Learning Enhancement in Healthy Young Adults
Brief Title: Effect of Number of Remote Limb Ischemic Conditioning Cycles on Learning Enhancement
Acronym: RLICC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Catherine E. Lang, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIHR01HD085930-Aim2; R01HD085930 (NIH)
Record Dates: First submitted 2018-04-18; First posted 2018-04-30 (Actual); Results first posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Healthy, Young Adults
Keywords: ischemic conditioning, motor learning

STUDY DESIGN:
Intervention Model Description: Single blinded, randomized controlled trial
Who Masked: Participant
Masking Description: Participants will be masked to their group assignment (RLIC or Sham conditioning) throughout the study. Participants will intuitively know the dose (number of cycles) of their assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RLIC - 5 Cycles (Experimental): Remote Limb Ischemic Conditioning (RLIC) is achieved via blood pressure cuff inflation to 20 mmHg above systolic blood pressure on the non-dominant arm. 5 Cycles of RLIC requires 45 minutes and involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. RLIC is performed on visits 1-7.
  Interventions: Behavioral: RLIC - 5 cycles; Behavioral: Balance training; Behavioral: Arm training; Behavioral: Sequence production training
- RLIC - 4 Cycles (Experimental): RLIC is achieved via blood pressure cuff inflation to 20 mmHg above systolic blood pressure on the non-dominant arm. 4 Cycles of RLIC requires 35 minutes and involves 4 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. RLIC is performed on visits 1-7.
  Interventions: Behavioral: RLIC - 4 Cycles; Behavioral: Balance training; Behavioral: Arm training; Behavioral: Sequence production training
- RLIC - 3 Cycles (Experimental): RLIC is achieved via blood pressure cuff inflation to 20 mmHg above systolic blood pressure on the non-dominant arm. 3 Cycles of RLIC requires 25 minutes and involves 3 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. RLIC is performed on visits 1-7.
  Interventions: Behavioral: RLIC - 3 Cycles; Behavioral: Balance training; Behavioral: Arm training; Behavioral: Sequence production training
- Sham Conditioning (Sham Comparator): Sham conditioning is achieved via blood pressure cuff inflation to 10 mmHg under diastolic blood pressure on the non-dominant arm. Sham conditioning requires 45 minutes and involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. Sham conditioning is performed on visits 1-7.
  Interventions: Behavioral: Sham conditioning; Behavioral: Balance training; Behavioral: Arm training; Behavioral: Sequence production training

INTERVENTIONS:
Behavioral: RLIC - 5 cycles — RLIC is achieved as listed in the arm/group descriptions. RLIC is performed on visits 1-7, which occur on consecutive weekdays.
  Other Names: Ischemic conditioning
  Arms: RLIC - 5 Cycles
Behavioral: RLIC - 4 Cycles — RLIC is achieved as listed in the arm/group descriptions. RLIC is performed on visits 1-7, which occur on consecutive weekdays.
  Other Names: Ischemic conditioning
  Arms: RLIC - 4 Cycles
Behavioral: RLIC - 3 Cycles — RLIC is achieved as listed in the arm/group descriptions. RLIC is performed on visits 1-7, which occur on consecutive weekdays.
  Other Names: Ischemic conditioning
  Arms: RLIC - 3 Cycles
Behavioral: Sham conditioning — Sham conditioning is achieved as listed in the arm/group descriptions. Sham conditioning is performed on visits 1-7, which occur on consecutive weekdays.
  Arms: Sham Conditioning
Behavioral: Balance training — All participants undergo training on a balance board, learning to hold the board level with equal weight on each leg. Participants perform the balance task for 15, 30-second trials per day at visits 3-7.
Behavioral: Arm training — All participants undergo training on a cup stacking task, learning to assemble and disassemble cup configurations as fast as they can. Participants perform the cup stacking task 5 trials per day at visits 3-7.
  Other Names: Cup stacking
Behavioral: Sequence production training — All participants undergo training on a discrete sequence production task. Participants learn to associate specific color and shape symbols with sequences of key presses on a keyboard. Participants perform the sequence production task for 10-15 minutes per day at visits 3-7.

SUMMARY:
The purpose of this research study is to determine the effect of number of remote limb ischemic conditioning (RLIC) cycles on enhancing learning in neurologically intact young adults.

DETAILED DESCRIPTION:
It is now understood that the nervous system has remarkable adaptive capacity. Specifically, the central nervous system retains its ability to reorganize in structure and function in response to behavioral experience in neurologically intact people and in individuals with neurological injury. Cognitive and motor learning guide the adaptation of the central nervous system and are essential components of effective training paradigms.

There is a growing body of literature which suggests that inducing a transient state of systemic ischemia has the potential to induce spinal plasticity, strengthen spared pathways to motorneurons, and lead to improved motor recovery following neurological injury.1,2 Specifically, daily systemic ischemic conditioning has been shown to improve both forelimb and respiratory motor function in rodent models of chronic cervical spinal injury.1,3 Moreover, systemic ischemic conditioning resulted in increased ankle strength (single session)2 and augmented walking speed and endurance (5 sessions)4 in humans with motor incomplete spinal cord injuries.

In a related area of research, it has been shown that ischemic conditioning administered peripherally represents a strategy for harnessing the body's endogenous protective capabilities against lethal levels of ischemia. With this technique, applying brief ischemia and reperfusion to a remote organ or tissue results in significantly reduced damage from subsequent exposures to ischemia. For example, applying a tourniquet and creating hypoxia in a rat's hindlimb for 10 minutes reduced the extent of cardiac abnormalities following a sustained ischemic insult.5 This same phenomenon has been shown in humans. Applying an inflated blood pressure cuff to the upper or lower limb has shown efficacy for protection in people undergoing cardiac surgeries,6,7 undergoing elective surgery to repair abdominal aortic aneurysm,8 experiencing MI,9 and with symptomatic intracranial arterial stenosis.7

The mechanisms underlying the neuroplastic and neuroprotective effects of ischemic conditioning are not fully understood. At this time, the literature indicates that there are both humoral and neural mechanisms responsible for the protection and the plasticity. It is clear that ischemic conditioning results in widespread physiological effects and that the observed effects work through multiple mechanistic pathways.

The next translational step is to investigate whether combining ischemic conditioning with behavioral training has the ability to augment motor learning. Specifically, we will employ remote limb ischemic conditioning (via inflation/deflation of a blood pressure cuff) with the objective of activating the endogenous pathways shown to elicit neuroplasticity. If eventually effective, RLIC could have profound effect on the rehabilitation and recovery of motor function in people with stroke. It is important to first start this translational investigation in neurologically intact people in order to determine optimal protocols for people with stroke.

The purpose of this study is to test the effect of number of RLIC cycles on motor learning in neurologically intact adults and if we can find a physiological blood marker related to effective administration of RLIC. We hypothesize that 3 cycles of RLIC will be sufficient to enhance motor leaning compared to sham conditioning, and that there will be a dose-dependent (number of cycles) response in learning, thus making training more efficient, more effective, and longer-lasting. Determining the number of cycles necessary to elicit the benefits of RLIC is important in developing the most effective and least burdensome treatment for future patients with motor deficits.

ELIGIBILITY:
Inclusion Criteria:

1. Between the age of 18 and 40 years

Exclusion Criteria:

1. History of neurological condition (i.e. stroke, Alzheimer's disease, Parkinson's disease), ADD, ADHD, balance impairment, or vestibular disorder
2. History of sleep apnea
3. History of lower extremity condition, injury, or surgery which could compromise performance on motor training task
4. Any extremity soft tissue, orthopedic, or vascular injury (i.e. peripheral vascular disease) which may contraindicate RLIC
5. Any cognitive, sensory, or communication problem that would prevent completion of the study
6. Current intensive weight lifting or interval training exercise
7. Current substance abuse or dependence
8. Current use of medication with selective serotonin-reuptake inhibitors.
9. Unwillingness to travel for all study visits

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lang, PT, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, all of the individual participant data after de-identification will be submitted to Washington University data repository.
Supporting Information: Study Protocol, SAP
Time Frame: Following publication
Access Criteria: Data will be available to anyone who wishes to access it through Washington University data repository.
URL: https://openscholarship.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- RLIC - 5 Cycles: Remote Limb Ischemic Conditioning (RLIC) is achieved via blood pressure cuff inflation on the non-dominant arm. 5 Cycles of RLIC requires 45 minutes and involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. RLIC is performed on visits 1-7.
  RLIC - 5 cycles: RLIC is achieved as listed in the arm/group descriptions. RLIC is performed on visits 1-7, which occur on consecutive weekdays.
  Balance training: All participants undergo training on a balance board, learning to hold the board level with equal weight on each leg. Participants perform the balance task for 15, 30-second trials per day at visits 3-7.
  Arm training: All participants undergo training on a cup stacking task, learning to assemble and disassemble cup configurations as fast as they can. Participants perform the cup stacking task 5 trials per day at visits 3-7.
  Sequence production training: All participants underg
- RLIC - 4 Cycles: RLIC is achieved via blood pressure cuff inflation on the non-dominant arm. 4 Cycles of RLIC requires 35 minutes and involves 4 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. RLIC is performed on visits 1-7.
  RLIC - 4 Cycles: RLIC is achieved as listed in the arm/group descriptions. RLIC is performed on visits 1-7, which occur on consecutive weekdays.
  Balance training: All participants undergo training on a balance board, learning to hold the board level with equal weight on each leg. Participants perform the balance task for 15, 30-second trials per day at visits 3-7.
  Arm training: All participants undergo training on a cup stacking task, learning to assemble and disassemble cup configurations as fast as they can. Participants perform the cup stacking task 5 trials per day at visits 3-7.
  Sequence production training: All participants undergo training on a discrete sequence pr
- RLIC - 3 Cycles: RLIC is achieved via blood pressure cuff inflation on the non-dominant arm. 3 Cycles of RLIC requires 25 minutes and involves 3 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. RLIC is performed on visits 1-7.
  RLIC - 3 Cycles: RLIC is achieved as listed in the arm/group descriptions. RLIC is performed on visits 1-7, which occur on consecutive weekdays.
  Balance training: All participants undergo training on a balance board, learning to hold the board level with equal weight on each leg. Participants perform the balance task for 15, 30-second trials per day at visits 3-7.
  Arm training: All participants undergo training on a cup stacking task, learning to assemble and disassemble cup configurations as fast as they can. Participants perform the cup stacking task 5 trials per day at visits 3-7.
  Sequence production training: All participants undergo training on a discrete sequence pr
- Sham Conditioning: Sham conditioning is achieved via blood pressure cuff inflation to 10 mmHg under diastolic blood pressure on the non-dominant arm. Sham conditioning requires 45 minutes and involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. Sham conditioning is performed on visits 1-7.
  Sham conditioning: Sham conditioning is achieved as listed in the arm/group descriptions. Sham conditioning is performed on visits 1-7, which occur on consecutive weekdays.
  Balance training: All participants undergo training on a balance board, learning to hold the board level with equal weight on each leg. Participants perform the balance task for 15, 30-second trials per day at visits 3-7.
  Arm training: All participants undergo training on a cup stacking task, learning to assemble and disassemble cup configurations as fast as they can. Participants perform the cup stacking task 5 trials per day at visits 3-7.
  Sequence production training: All
Period: Overall Study
Arm/Group | RLIC - 5 Cycles | RLIC - 4 Cycles | RLIC - 3 Cycles | Sham Conditioning
Started | 10 | 10 | 11 | 9
Completed | 10 | 10 | 11 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RLIC - 5 Cycles | RLIC - 4 Cycles | RLIC - 3 Cycles | Sham Conditioning | Total
Number analyzed (Participants) | 10 | 10 | 11 | 9 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (3.9) | 25.9 (2.9) | 26.2 (4.6) | 26.1 (1.6) | 25.9 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 6 | 8 | 28
  Male | 3 | 3 | 5 | 1 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 3 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 1 | 7
  White | 6 | 7 | 6 | 5 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 11 | 9 | 40
Body Mass Index [Mean (Standard Deviation); unit: kg/m*m] | 24.1 (6.6) | 23.9 (4.3) | 26.7 (5.3) | 27.2 (8.1) | 25.5 (6.1)
Resting systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 113 (14) | 116 (14) | 117 (11) | 116 (12) | 116 (13)
Resting diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 73 (10) | 74 (10) | 75 (8) | 74 (8) | 74 (9)

OUTCOME MEASURES:

1. Primary Outcome: Balance Score
Description: The change from Visit 1 to Visit 7 in the average amount of time in seconds that a participant maintains the stability platform within ±3° of horizontal position during 5 trials of 30 seconds each. A greater increase in the balance score means more learning has occurred over the course of the study.
Time Frame: Visit 1 and Visit 7, approximately 1 week
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | RLIC - 5 Cycles | RLIC - 4 Cycles | RLIC - 3 Cycles | Sham Conditioning
Number analyzed (Participants) | 10 | 10 | 11 | 9
seconds | 9.9 (4.6) | 11.5 (5.7) | 7.0 (5.1) | 11.3 (4.6)
Statistical Analysis 1: Comparison: RLIC - 5 Cycles vs RLIC - 4 Cycles vs RLIC - 3 Cycles vs Sham Conditioning; Test type: Superiority; p = 0.172, ANOVA

2. Primary Outcome: Cup Stacking Score
Description: The change from Visit 1 to Visit 7 in the average amount of time in seconds that a participant takes to stack and unstack pre-determined patterns of cups. A greater decrease in the cup stacking score means more learning has occurred over the course of the study.
Time Frame: Visit 1 and Visit 7, approximately 1 week
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | RLIC - 5 Cycles | RLIC - 4 Cycles | RLIC - 3 Cycles | Sham Conditioning
Number analyzed (Participants) | 10 | 10 | 11 | 9
seconds | -22.2 (8.8) | -14.9 (3.5) | -11.9 (10.4) | -10.1 (14.8)
Statistical Analysis 1: Comparison: RLIC - 5 Cycles vs RLIC - 4 Cycles vs RLIC - 3 Cycles vs Sham Conditioning; Test type: Superiority; p = 0.169, ANOVA

3. Primary Outcome: Discrete Sequence Production Task Score
Description: The change from Visit 1 to Visit 7 in the average amount of time in seconds that a participant takes to complete pre-determined patterns of keypresses. A greater decrease in the Discrete Sequence Production Task score means more learning has occurred over the course of the study.
Time Frame: Visit 1 and Visit 7, approximately 1 week
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | RLIC - 5 Cycles | RLIC - 4 Cycles | RLIC - 3 Cycles | Sham Conditioning
Number analyzed (Participants) | 10 | 10 | 11 | 9
seconds | -3.1 (0.7) | -2.9 (0.3) | -2.6 (0.6) | -2.9 (0.3)
Statistical Analysis 1: Comparison: RLIC - 5 Cycles vs RLIC - 4 Cycles vs RLIC - 3 Cycles vs Sham Conditioning; Test type: Superiority; p = 0.501, ANOVA

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | RLIC - 5 Cycles | RLIC - 4 Cycles | RLIC - 3 Cycles | Sham Conditioning
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT03512041/Prot_SAP_000.pdf